CLINICAL TRIAL: NCT00006306
Title: Effects of Chronic Ozone Exposure on Lung Function
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 134; R01HL060689 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2006-01

CONDITIONS: Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To determine the effects of chronic ozone exposure on lung function in young men and women.

DETAILED DESCRIPTION:
BACKGROUND:

A large part of the U.S. population is exposed to ambient ozone (O3) concentrations that are associated with acute respiratory health effects; however, little is known about the effects on human respiratory health of long-term exposure to such ambient concentrations. Chronic exposure of non-human primates to high concentrations of O3 are associated with pathologic changes in the centriacinar region of the lung that are similar to changes observed in young cigarette smokers. This is the first detailed epidemiologic study of the effects of chronic exposure to an air pollutant based on individual estimates of lifetime exposure and controlled exposure data. The study tests a specific toxicologic model in humans that has relevance for chronic respiratory disease and explores mechanisms of effects.

DESIGN NARRATIVE:

The study tested the hypothesis that, in humans, there was an exposure-response relationship between the amount of chronic exposure to ambient O3 and measures of lung function that reflected changes in the centriacinar region of the human lung (FEF25-75); and this relationship was not seen with measures of more proximal airway function (FEV1). First-year UC Berkeley students, ages 18-21 yrs, who were lifelong residents of the Los Angles Basin, (high O3) and the San Francisco Bay Area, (low O3) were studied. Lifetime exposure to ambient O3 was estimated with methods developed by the investigators that combined questionnaire and ambient O3 data. Lung function was assessed with maximum expiratory flow-volume curves. Students were studied after 4-6 months of low ambient O3 exposure and immediately after 2-3 months of exposure to summertime O3. Students from each area who were at the upper and lower tails of the FEF25-75 distribution underwent two controlled O3 exposures (seasonal as above) followed by bronchoalveolar lavage/biopsy to evaluate relationships between measures of inflammation, injury/repair and oxidant induced damage/repair and FEF25-75. Regression was used to evaluate relationships between lifetime O3 exposure and lung function, adjusted for past and family respiratory history, allergy history, home characteristics, exposure to environmental tobacco smoke and particle air pollution and NO2.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Tager — University of California, Berkeley

REFERENCES:
- [Background] Tager IB, Balmes J, Lurmann F, Ngo L, Alcorn S, Kunzli N. Chronic exposure to ambient ozone and lung function in young adults. Epidemiology. 2005 Nov;16(6):751-9. doi: 10.1097/01.ede.0000183166.68809.b0. PMID 16222164